CLINICAL TRIAL: NCT03303131
Title: Discharge From Community-based Management of Severe Acute Malnutrition Using Mid Upper Arm Circumference
Brief Title: SAM: Discharge Based on the Use of a MUAC-based Criterion to
Status: Completed | Type: Observational
Sponsor: Epicentre (Other)
Collaborators: Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Sponsor
Other Study IDs: MUAC 2007-2011
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Severe Acute Malnutrition
MeSH Terms: conditions — Severe Acute Malnutrition

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Period A: Children discharged as recovered from September 2007 to March 2009 with at least 15% of their weight at admission
  Interventions: Other: Discharge from community-based management
- Period B: Children discharged as recovered from April 2009 to December 2011 with Children discharged as recovered from September 2007-March 2009 with MUAC ≥ 124 mm
  Interventions: Other: Discharge from community-based management

INTERVENTIONS:
Other: Discharge from community-based management — Comparison of patient characteristics and treatment outcomes between two groups

SUMMARY:
Retrospective analysis of routine program data of children aged 6 to 59 months admitted to the MSF therapeutic feeding program with MUAC ≤ 118 mm in Yako and Titao districts of Burkina Faso from 2007-2011.

DETAILED DESCRIPTION:
Comparison of patient characteristics and treatment outcomes was conducted between two groups: 1) children discharged as recovered from September 2007 to March 2009 with at least 15% of their weight at admission (Period A); and 2) children discharged as recovered from April 2009 to December 2011 with MUAC ≥ 124 mm (Period B).

A total of 50,841 children were admitted with MUAC ≤ 118 mm to the MSF therapeutic feeding program and were included in this analysis: 24,792 children in Period A (2007-2009) and 26,049 children in Period B (2009-2011).

Overall, 89% of admissions were directly into outpatient care and the majority (53%) entered with a MUAC 116-118mm; 48% of children were male and 80% of children < 2 years of age (Table 1).

Compared to children admitted in Period A, children admitted in Period B were statistically more likely to be female, younger, and of better anthropometric status (e.g. higher mean MUAC, WHZ and HAZ).

There was a greater proportion of children admitted directly to inpatient care in Period B than in Period A (10.6% vs 8.0%).

ELIGIBILITY:
Inclusion Criteria:

* 6 to 59 months old
* presence of bipedal pitting edema or MUAC ≤ 118 mm

Exclusion Criteria:

* < 6 months old or > 59 months old
* absence of bipedal pitting edema or MUAC ≥ 118 mm

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children admitted to the MSF therapeutic feeding program in Yako and Titao districts from September 2007 to December 2011
Sampling Method: Non-Probability Sample
Enrollment: 50841 (Actual)
Dates: Start 2007-09-01 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2011-12-31 (Actual)

PRIMARY OUTCOMES:
MUAC based criterion | 52 months
  Use of a discharge criterion of MUAC ≥ 124 mm

IPD SHARING:
Plan to Share IPD: No